CLINICAL TRIAL: NCT00916071
Title: Association Between Attention Deficit Hyperactivity Disorder and Bulimia Nervosa in Outpatients With Eating Disorders
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Hilda and Preston Davis Foundation (Unknown)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Scientific Coordinator of the Adult ADHD Program, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2007-P-002374
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-01

CONDITIONS: Bulimia Nervosa; Eating Disorders; ADHD
Keywords: Bulimia Nervosa; Eating Disorder NOS; Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eating Disorders: Study subjects will be individuals with a history of eating disorder(s) diagnosis

SUMMARY:
To understand whether a relationship exists between eating disorders and ADHD, we seek to clarify the prevalence of ADHD in individuals with eating disorders. To this end, we will estimate the prevalence of ADHD, and other neuropsychiatric disorders, in outpatients with history of an eating disorder diagnosis. Secondarily, we will identify patterns of cognitive deficits in outpatients with history of an eating disorder diagnosis. We will also examine whether ADHD in this population is associated with functional and familial correlates associated with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between, and including, 18 and 55 years of age with a history of eating disorder diagnosis.

Exclusion Criteria:

* Any clinically unstable psychiatric conditions such as: acute psychosis, acute panic, acute obsessive compulsive disorder, acute mania, acute suicidality, acute substance use disorders (alcohol or drugs), and sociopathy.
* Any metabolic, neurological, hepatic, renal, cardiovascular, hematological, opthalmic, or endocrine disease that would confound ability to participate in valid assessments.
* Mental retardation (IQ <75).
* Organic brain disorders.
* Non-English speaking subjects will not be allowed into the study because the assessment instruments are unavailable and have not been adequately standardized in other languages.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male and female outpatients between, and including, 18 and 55 years of age with a history of eating disorder diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
We will identify the lifetime rate of mental health conditions using structured clinical interviews in subjects with a lifetime history of eating disorders and compare the rate of these conditions to that of non-ED control subjects. | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital